CLINICAL TRIAL: NCT04774731
Title: A Randomized Controlled Trial to Evaluate the Efficacy of Whole Body Vibration on Walking Performance in Elderly Hemodialysis Patients
Brief Title: Effect of Whole Body Vibration on Walking Performance in Elderly Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osaka University (Other)
Responsible Party: Principal Investigator, Yusuke Sakaguchi, assistant professor, Osaka University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WBV-HD
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Hemodialysis
Keywords: whole body vibration; hemodialysis; gait function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole Body Vibration (Experimental)
  Interventions: Other: Whole Body Vibration
- Control (No Intervention)

INTERVENTIONS:
Other: Whole Body Vibration — Receiving WBV training three times a week before initiation of dialysis sessions for 12 weeks. Subjects stand on a platform of WBV for 3 minutes in every training session.
  Arms: Whole Body Vibration

SUMMARY:
The purpose of this study is to evaluate the efficacy of whole body vibration for 12 weeks on walking performance in elderly hemodialysis patients.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized controlled trial. Eligible subjects will be randomized in a 1:1 ratio to a whole-body vibration (WBV) group or controlled group. Patients in a WBV group will receive WBV training three times a week before initiation of dialysis sessions for 12 weeks. The primary outcome of the study will be the change in walking performance assessed by the timed up and go test.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing maintenance hemodialysis three times a week .

Exclusion Criteria:

* Having difficulty in walking by oneself.
* Having difficulty in receiving whole body vibration training because of cognitive impairment.
* History of fracture of lower limb within 1 year.
* History of total hip arthroplasty.
* Unsuitable for participant in the trial by an attending physician.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Change in the timed up and go test | 12 weeks after starting intervention

SECONDARY OUTCOMES:
Change in the one-leg standing test | 12 weeks after starting intervention
Change in the 30-second chair-stand test | 12 weeks after starting intervention

CONTACTS AND LOCATIONS:
Overall Officials: Yusuke Sakaguchi, MD, PhD, Principal Investigator — Department of Nephrology, Osaka University
Locations (1):
- Osaka University Hospital, Suita, Osaka, Japan

REFERENCES:
- [Derived] Asahina Y, Sakaguchi Y, Kajimoto S, Hattori K, Oka T, Kaimori JY, Kashihara N, Isaka Y. A Randomized Controlled Trial of Whole-Body Vibration on Gait Ability and Balance among Older Hemodialysis Patients. Clin J Am Soc Nephrol. 2023 Jan 1;18(1):84-90. doi: 10.2215/CJN.0000000000000018. PMID 36719160